CLINICAL TRIAL: NCT02189980
Title: Aromatherapy Using a Nasal Clip After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Balanced Health plus (Industry)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BHp2014-001
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Post-operative Nausea
Keywords: Nausea; Post-operative
MeSH Terms: conditions — Nausea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saline & nasal clip (Placebo Comparator): Saline and nasal clip inhaled post-operatively
  Interventions: Other: Duration of effectiveness of the essential oil blend; Other: Participant comfort using the nasal clip delivery system
- Aromatherapy blend & nasal clip (Experimental): Aromatherapy blend and nasal clip inhaled post-operatively
  Interventions: Other: Aromatherapy blend; Other: Duration of effectiveness of the essential oil blend; Other: Participant comfort using the nasal clip delivery system

INTERVENTIONS:
Other: Aromatherapy blend — A blend of 45% ginger, 25% peppermint, 5% spearmint, and 25% cardamom essential oils
  Arms: Aromatherapy blend & nasal clip
Other: Duration of effectiveness of the essential oil blend — Evidence of effectiveness of tested aromatherapy blend in reducing symptoms of post-operative nausea as measured by patient self-report using Likert-type scale measure immediately to one-day post-operative.
Other: Participant comfort using the nasal clip delivery system — Comfort of participants using nasal clip delivery system for aromatherapy will be measured by self-report using Likert-type scale immediately to one-day post-operative.

SUMMARY:
The purpose of this follow up study is to determine the duration of action regarding aromatherapy to treat nausea occurring postoperatively.

DETAILED DESCRIPTION:
The primary hypothesis of the study is that post-operative patients who meet eligibility criteria and report nausea and receive a blend of 45% ginger, 25% peppermint, 5% spearmint, and 25% cardamom essential oils while using a nasal clip to facilitate inhalation will have more relief from nausea than those who receive normal saline inhalation using the same delivery system.

The secondary purposes of the study is to determine the duration of effectiveness of the essential oil blend as compared to the saline in the relief of post-operative nausea and to investigate the degree of comfort participants report using the nasal clip delivery system for aromatherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* cognitively able to give consent based on nurse's assessment,
* having gynecological or other abdominal surgery
* not allergic to peppermint, spearmint, cardamom or ginger
* not receiving blood thinning medications

Exclusion Criteria:

* less than 18 years old
* unable to cognitively give consent
* allergic to ginger, peppermint, cardamom or spearmint.
* receiving warfarin (Coumadin) or any antiplatelet drug (heparin, 325 mg Aspirin, clopidogrel (Plavix) or other) or a diagnosis of bleeding diatheses (predisposition to abnormal blood clotting/hemorrhage) will not be included in this study.
* all surgeries other than gynecological or abdominal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Duration of effectiveness of the essential oil blend | Immediately to one-day post-operative
  Evidence of effectiveness of tested aromatherapy blend in reducing symptoms of post-operative nausea as measured by patient self-report using Likert-type scale measure.

SECONDARY OUTCOMES:
Participant comfort using the nasal clip delivery system | Immediately post-op to one-day post-op
  Comfort of participants using nasal clip delivery system for aromatherapy will be measured by self-report using Likert-type scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hunt, MD, Principal Investigator — Balanced Health plus
Locations (1):
- CMC -- University, Charlotte, North Carolina, United States